CLINICAL TRIAL: NCT00053352
Title: A Phase III Study Of Reduced Therapy In The Treatment Of Children With Low And Intermediate Risk Extracranial Germ Cell Tumors
Brief Title: Surgery and Combination Chemotherapy in Treating Children With Extracranial Germ Cell Tumors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGCT0132; NCI-2009-00373 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000269433 (Other: Clinical Trials.gov); COG-AGCT0132 (Other: Children's Oncology Group); U10CA098543 (NIH)
Record Dates: First submitted 2003-01-27; First posted 2003-01-28 (Estimated); Results first posted 2017-12-08 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Childhood Embryonal Tumor; Childhood Extracranial Germ Cell Tumor; Childhood Extragonadal Germ Cell Tumor; Childhood Malignant Ovarian Germ Cell Tumor; Childhood Malignant Testicular Germ Cell Tumor; Childhood Teratoma; Ovarian Embryonal Carcinoma; Ovarian Yolk Sac Tumor; Stage II Malignant Testicular Germ Cell Tumor; Stage IIA Ovarian Germ Cell Tumor; Stage IIB Ovarian Germ Cell Tumor; Stage IIC Ovarian Germ Cell Tumor; Stage III Malignant Testicular Germ Cell Tumor; Stage IIIA Ovarian Germ Cell Tumor; Stage IIIB Ovarian Germ Cell Tumor; Stage IIIC Ovarian Germ Cell Tumor; Testicular Choriocarcinoma and Yolk Sac Tumor; Testicular Embryonal Carcinoma
MeSH Terms: conditions — Ovarian Germ Cell Cancer; Testicular Neoplasms; Teratoma; Endodermal Sinus Tumor | interventions — Surgical Procedures, Operative; Congresses as Topic; Cisplatin; Etoposide; Bleomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients enrolled with gonadal tumors of stage II or greater or extragonadal tumors of any stage receive cisplatin IV over 90 minutes & etoposide IV over 90 minutes days 1-3 and bleomycin sulfate IV over ≥ 10 minutes day 1. Treatment repeats every 3 weeks, 3 courses (weeks 0,3 & 6).
  After completion of compressed induction chemotherapy, patients with no change in disease status or disease progression are removed from study. Patients with no evidence of disease receive no further therapy. Patients with a partial response or abnormal tumor markers proceed to conventional surgery (second-look) and/or 3 more courses of compressed consolidation chemotherapy.
  After surgery, patients with pathologic complete response and have normal tumor markers receive no further therapy. Patients who remain with a partial response after surgery receive compressed consolidation chemotherapy.
  Patients receive cisplatin, etoposide, and bleomycin as induction chemotherapy in weeks 10,13, & 16.
  Interventions: Procedure: conventional surgery; Drug: cisplatin; Drug: etoposide; Biological: bleomycin sulfate; Other: laboratory biomarker analysis
- Arm 2 (No Intervention): Patients who are enrolled with stage I gonadal tumors receive no further anticancer therapy until evidence of tumor recurrence or the diagnosis of a second malignant neoplasm.
  Observation only for recurrence or development of an SMN

INTERVENTIONS:
Procedure: conventional surgery
  Other Names: surgery, conventional
  Arms: Arm I
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
  Arms: Arm I
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
  Arms: Arm I
Biological: bleomycin sulfate — Given IV
  Other Names: Blenoxane; BLEO; BLM
  Arms: Arm I
Other: laboratory biomarker analysis — Correlative studies
  Arms: Arm I

SUMMARY:
This phase III trial is studying surgery followed by combination chemotherapy to see how well it works in treating children with germ cell tumors that are not located in the head. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug, and giving them after surgery, may kill any remaining tumor cells following surgery. It is not yet known whether combination chemotherapy is effective in decreasing the recurrence of childhood germ cell tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine whether children with newly diagnosed low- or intermediate-risk extracranial germ cell tumors (GCTs) can maintain a 3-year event-free survival of at least 92% (for intermediate-risk tumors only) and overall survival of at least 95% (both low-risk and intermediate-risk tumors) after treatment with surgery followed by compressed cisplatin, etoposide, and bleomycin (low-risk disease closed to accrual as of 01/20/10).

II. Determine the percentage of patients with stage I ovarian or stage I testicular GCTs for whom chemotherapy can be eliminated.

III. Determine the percentage of intermediate-risk patients who require only 3 courses of therapy.

IV. Determine the acute toxic effects of compressed therapy in these patients. V. Determine the long-term sequelae in patients treated with this regimen. VI. Determine the number of hospital days and total drug doses required for patients treated with compressed therapy.

VII. Compare the number of protocol-directed treatment days used in CCG-8882 vs the number of treatment days used in this study.

VIII. Determine the cytogenetic and molecular genetic features in patients treated with this regimen.

OUTLINE: Patients are stratified according to disease risk (low vs intermediate).

SURGERY: Patients undergo surgical resection.

Low-risk disease: Patients with gonadal primaries and no evidence of disease after surgery undergo monitoring for disease progression. Patients who remain disease free receive no further treatment. Patients who have disease progression after surgery receive compressed induction chemotherapy. (closed to accrual as of 01/20/2010)

Intermediate-risk disease: After surgery, patients proceed to compressed induction chemotherapy.

COMPRESSED INDUCTION CHEMOTHERAPY: Patients receive cisplatin IV over 90 minutes and etoposide IV over 90 minutes on days 1-3 and bleomycin IV over ≥ 10 minutes on day 1. Treatment repeats every 3 weeks for 3 courses (weeks 0, 3, and 6).

After completion of compressed induction chemotherapy, patients who have no change in disease status or disease progression are removed from study. Patients with no evidence of disease receive no further therapy. Patients with a partial response or who have abnormal tumor markers proceed to second-look surgery and/or 3 more courses of compressed consolidation chemotherapy.

SECOND-LOOK SURGERY: Patients undergo surgical resection of residual tumor. After surgery, patients who are in pathologic complete response and have normal tumor markers receive no further therapy. Patients who remain with a partial response after surgery receive compressed consolidation chemotherapy.

COMPRESSED CONSOLIDATION CHEMOTHERAPY: Patients receive cisplatin, etoposide, and bleomycin as in induction chemotherapy in weeks 10, 13, and 16.

Patients are followed up monthly for 6 months, every 3 months for 18 months, and then annually for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Extracranial germ cell tumor that contains 1 of the following malignant histologies: NOTE: Mixed germ cell tumors that include mature/immature teratoma are eligible provided 1 of the 3 histologies listed above is also present in the tumor.

  * Yolk sac tumor
  * Embryonal carcinoma
  * Choriocarcinoma
* Low-risk disease (closed to accrual as of 01/20/10)

  * Stage I gonadal tumors (ovarian and testicular)
  * Must have undergone complete surgical and radiologic staging to exclude the possibility of > stage I disease
* Intermediate-risk disease

  * Stage II, III, or IV malignant testicular GCT
  * Stage II or III malignant ovarian GCT
  * Stage I or II malignant extragonadal GCT
  * Previously stage I gonadal patients who have relapsed on the low-risk (observation) stratum of this study(closed to accrual as of 01/20/10)
  * Patients with immature teratoma or mature teratoma who relapse with a malignant component
* No patients with any of the following diagnoses:

  * Stage IV ovarian and stage III-IV extragonadal GCT
  * Intracranial GCT
  * Pure mature or immature teratoma, pure dysgerminoma, or seminoma
  * Patients with a non-germ cell component in their GCT (e.g., primitive neuroectodermal tumors or rhabdomyosarcoma)
* Alpha-fetoprotein and beta human chorionic gonadotropin tumor markers known

  * If > 5 days have elapsed from the time of obtaining original markers, tumor markers must be repeated before enrollment of low-risk patients and before initiating therapy in intermediate-risk patients (the results of the repeated tumor markers do not have to be known at the time of study enrollment)
* Must be enrolled within 6 weeks of original diagnostic surgery
* Creatinine clearance or radioisotope GFR ≥ 70 mL/min OR a serum creatinine based on age/gender as follows:

  * ≤ 0.4 mg/dL (for patients 1 to 5 months of age)
  * ≤ 0.5 mg/dL (for patients 6 to 11 months of age)
  * ≤ 0.6 mg/dL (for patients 1 year of age)
  * ≤ 0.8 mg/dL (for patients 2 to 5 years of age)
  * ≤ 1.0 mg/dL (for patients 6 to 9 years of age)
  * ≤ 1.2 mg/dL (for patients 10 to 12 years of age)
  * ≤ 1.4 mg/dL (for female patients ≥ 13 years of age)
  * ≤ 1.5 mg/dL (for male patients 13 to 15 years of age)
  * ≤ 1.7 mg/dL (for male patients ≥ 16 years of age)
* No prior chemotherapy
* No prior radiotherapy

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 302 (Actual)
Dates: Start 2003-11-03 (Actual); Primary Completion 2013-10-01 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Frazier, MD, Principal Investigator — Children's Oncology Group
Locations (126):
- United States (112):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's Hospital, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Childrens Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Sutter General Hospital, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - University of California San Francisco Medical Center-Parnassus, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Lee Memorial Health System, Fort Myers, Florida
  - University of Florida, Gainesville, Florida
  - Memorial Healthcare System - Joe DiMaggio Children's Hospital, Hollywood, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - University of Hawaii, Honolulu, Hawaii
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Childrens Memorial Hospital, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Hope Children's Hospital, Oak Lawn, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University, Springfield, Illinois
  - University of Kentucky, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Michigan State University - Breslin Cancer Center, Lansing, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Medical Center-Fairview, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - The Childrens Mercy Hospital, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - UMDNJ - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Albany Medical Center, Albany, New York
  - Brooklyn Hospital Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - New York University Langone Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospitals Inc, Asheville, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Medical Center-Fargo, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Children's Medical Center of Dayton, Dayton, Ohio
  - Mercy Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Hershey Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Palmetto Health Richland, Columbia, South Carolina
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Science Center-Amarillo, Amarillo, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - University of Vermont, Burlington, Vermont
  - Childrens Hospital-King's Daughters, Norfolk, Virginia
  - Carilion Clinic Children's Hospital, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - West Virginia University Charleston, Charleston, West Virginia
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (2):
  - The Children's Hospital at Westmead, Sydney, New South Wales
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (9):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Chedoke-McMaster Hospitals, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Hospital Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Ste-Foy, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
- Starship Children's Hospital, Grafton, Auckland, New Zealand
- San Jorge Children's Hospital, Santurce, Puerto Rico
- Swiss Pediatric Oncology Group - Geneva, Geneva, Switzerland

REFERENCES:
- [Derived] O'Neill AF, Xia C, Krailo MD, Shaikh F, Pashankar FD, Billmire DF, Olson TA, Amatruda JF, Villaluna D, Huang L, Malogolowkin M, Rodriguez-Galindo C, Frazier AL. alpha-Fetoprotein as a predictor of outcome for children with germ cell tumors: A report from the Malignant Germ Cell International Consortium. Cancer. 2019 Oct 15;125(20):3649-3656. doi: 10.1002/cncr.32363. Epub 2019 Jul 29. PMID 31355926
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I: Experimental
- Arm 2: No intervention
Period: Overall Study
Arm/Group | Arm I | Arm 2
Started | 190 | 112
Completed | 169 | 102
Not Completed | 21 | 10
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 11 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Ineligible | 8 | 8
Not completed — Disease at new site | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I | Arm 2 | Total
Number analyzed (Participants) | 190 | 112 | 302
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.57 (5.65) | 5.41 (5.93) | 8.02 (6.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 29 | 174
  Male | 45 | 83 | 128
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 14 | 10 | 24
  Native Hawaiian or Other Pacific Islander | 1 | 3 | 4
  Black or African American | 22 | 8 | 30
  White | 128 | 72 | 200
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 24 | 18 | 42
Region of Enrollment [Number; unit: participants]
  New Zealand | 2 | 3 | 5
  Canada | 16 | 8 | 24
  United States | 170 | 91 | 261
  Australia | 1 | 8 | 9
  Switzerland | 0 | 2 | 2
  Guam | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Event-Free Survival (EFS)
Description: Proportion of patients event free at 3 years following enrollment. Event-free survival is not a primary outcome measure for Arm 2 patients.
Time Frame: 3 Years after enrollment
Population: 181 patients were evaluated for event free survival through 3 years for patients enrolled on Arm 1. Event-free survival is not a primary outcome measure for Arm 2 patients.
Measure: Number (95% Confidence Interval); unit: Percent probability
Groups:
- Arm 1: Experimental
Arm/Group | Arm 1
Number analyzed (Participants) | 181
Percent probability | 87.0 [81.0 to 92.0]

2. Primary Outcome: Overall Survival (OS)
Description: Percentage probability of being alive at 3 years following enrollment.
Time Frame: 3 Years after enrollment
Measure: Number (95% Confidence Interval); unit: Percent Probability
Arm/Group | Arm I | Arm 2
Number analyzed (Participants) | 181 | 104
Percent Probability | 97.0 [93.0 to 99.0] | 99.0 [92.8 to 99.9]

3. Secondary Outcome: Days Hospitalized for Patients Who Receive Chemotherapy
Description: Calculated to quantify the treatment cost associated with this regimen.
Time Frame: Up to 126 days after the start of chemotherapy
Population: 182 patients were enrolled on intermediate risk chemotherapy and were evaluable for this secondary endpoint
Measure: Mean (Standard Deviation); unit: Days in the hospital
Arm/Group | Arm I
Number analyzed (Participants) | 182
Days in the hospital | 14.08 (10.27)

4. Secondary Outcome: Toxicity Associated With Chemotherapy: Grade 3 or Higher. Toxicity as Assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v4.0
Description: The number of patients assigned to receive chemotherapy that experience CTC Version 4 grade 3 or higher at any time during protocol therapy
Time Frame: Up to 126 days after the start of chemotherapy
Population: 182 patients were enrolled on intermediate risk chemotherapy and were evaluable for this secondary endpoint
Measure: Number; unit: patients
Arm/Group | Arm I
Number analyzed (Participants) | 182
patients
  Abdominal pain | 3
  Acute kidney injury | 1
  Lymphocyte count decrease | 2
  Iincrease in alanine aminotransferase | 1
  Neutrophil count decrease | 58
  Anemia | 10
  Increase in aspartate aminotransferase | 1
  Catheter related infection | 1
  Constipation | 1
  Dehydration | 1
  Encephalopathy | 1
  Febrile neutropenia | 9
  Fever | 3
  Hyperglycemia | 1
  Hyperkalemia | 1
  Hypocalcemia | 2
  Hypokalemia | 1
  Hypomagnesemia | 1
  Hyponatremia | 1
  Hypophosphatemia | 6
  Small intestine obstruction | 1
  Nausea | 5
  Non-cardiac chest pain | 1
  Other gastrointestinal disorders | 1
  Other infection | 10
  Platelet count decrease | 7
  Syncope | 1
  Vomiting | 4
  White blood cell decrease | 17
  Wound infection | 1

ADVERSE EVENTS:
Description: Only patients who are considered eligible contribute to the tabulation of adverse events. For Arm/Group Title "No Intervention" (Arm/Group Description: "Arm 2") 104 eligible patients contribute as described from the Participant Flow as 112 enrolled minus 8 ineligible. For Arm/Group Title "Experimental" (Arm/Group Description: "Arm 1") 182 eligible patients contribute as described from the Participant Flow as 190 enrolled minus 8 ineligible.
Groups:
- Arm 2 (Observation): Patients who are enrolled with stage I gonadal tumors receive no further anticancer therapy until evidence of tumor recurrence or the diagnosis of a second malignant neoplasm.
  Observation only for recurrence or development of an SMN
- Arm I (Chemotherapy): Patients enrolled with gonadal tumors of stage II or greater or extragonadal tumors of any stage receive cisplatin IV over 90 minutes & etoposide IV over 90 minutes days 1-3 and bleomycin sulfate IV over ≥ 10 minutes day 1. Treatment repeats every 3 weeks, 3 courses (weeks 0,3 & 6).
  After completion of compressed induction chemotherapy, patients with no change in disease status or disease progression are removed from study. Patients with no evidence of disease receive no further therapy. Patients with a partial response or abnormal tumor markers proceed to conventional surgery (2nd-look) and/or 3 more courses of compressed consolidation chemotherapy.
  After surgery, patients with pathologic complete response and have normal tumor markers receive no further therapy. Patients who remain with a partial response after surgery receive compressed consolidation chemotherapy.
  Patients receive cisplatin, etoposide, and bleomycin as induction chemotherapy in weeks 10,13, & 16.
  con
Arm/Group | Arm 2 (Observation) | Arm I (Chemotherapy)
Serious Adverse Events (participants affected / at risk) | 0/104 | 0/182
Other Adverse Events (participants affected / at risk) | 0/104 | 78/182
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 2 (Observation) (N=104) | Arm I (Chemotherapy) (N=182)
Abdominal pain (Gastrointestinal disorders) | 0 | 3
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 10
Aspartate aminotransferase increased (Investigations) | 0 | 1
Catheter related infection (Infections and infestations) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 9
Fever (General disorders) | 0 | 3
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 1
Hearing impaired (Ear and labyrinth disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 2
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 6
Ileus (Gastrointestinal disorders) | 0 | 0
Infections and infestations - Other, specify (Infections and infestations) | 0 | 10
Lymphocyte count decreased (Investigations) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 5
Neutrophil count decreased (Investigations) | 0 | 58
Non-cardiac chest pain (General disorders) | 0 | 1
Platelet count decreased (Investigations) | 0 | 7
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 4
White blood cell decreased (Investigations) | 0 | 17
Wound infection (Infections and infestations) | 0 | 1

LIMITATIONS AND CAVEATS:
Only patients considered eligible contribute to the tabulation of AEs. Arm 1: 182 eligible as described in Participant Flow as 190 enrolled, -8 ineligible. Arm 2: 104 eligible as described in Participant Flow as 112 enrolled, -8 ineligible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.